CLINICAL TRIAL: NCT03241381
Title: A Cross Sectional Observational Study
Brief Title: Prevalence of Serum-Vitamin D Abnormalities, Periodontitis and Anaemia in Patients With Melasma
Status: Completed | Type: Observational
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, NALLAN CHAITANYA, Associate Professor, department of oral medicine and radiology, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Other Study IDs: ECR/267/Indt/AP/2016
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Melasma, Periodontitis, Vitamin D Abnormalities, Anaemia
Keywords: observational sample
MeSH Terms: conditions — Melanosis; Periodontitis; Anemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A : Melasma: patients with facial pigmentation in the form of melasma
  Interventions: Diagnostic Test: vitamin D serum assay study and control groups; Diagnostic Test: Photometry; Other: Russels periodontal index
- Group B: Non Melasma: Patients without any facial pigmentation or melasma
  Interventions: Diagnostic Test: vitamin D serum assay study and control groups; Diagnostic Test: Photometry; Other: Russels periodontal index

INTERVENTIONS:
Diagnostic Test: vitamin D serum assay study and control groups — Serum- vitamin D assay
Diagnostic Test: Photometry — Serum- Hemoglobin assay
Other: Russels periodontal index — Clinical examination for periodontitis

SUMMARY:
Melasma is a commonly pigmention characterized by melanotic patches on the face. literature searched revealed that periodontitis and vitamin D deficiency have occurred along with anemia. Actinic associated factors may be indirectly related to vitamin D, melasma contributes to sun exposed area of face.To correlate melasma with clinical evidence of periodontitis and vitamin D serum analysis along side hb %. Patients with facial melasma between 30-70yrs of either gender formed Group A (95). Anaemia and periodontitis were Clinically checked. Additionally serum analysis of vitamin D and hb percentage were analysed. Similar procedure was carried out on controls which had Group B (95) patients with no melasma on face.

The study revealed significant correlation between melasma and periodontitis with vitamin D abnormalities (p value<.05), where as insignificant correlation between melasma and Hb%. The correlation between melasma, vitamin d changes and periodontitis may prompt the clinician to check for any such changes in any patient. Melasma in patients with periodontitis and serum vitamin D changes might be a considered as a syndrome.

DETAILED DESCRIPTION:
Melasma, is a relatively common chronic pigmentation of the face, although it may be localized also on the neck and forearms. It is also called as chloasma or mask of pregnancy. It has higher prevalence in women and occurs less commonly in men. It most commonly affects the sun-exposed areas of skin of face. Three patterns of presentation have been reported: Centro-facial, malar and mandibular forms. The interplay of various risk factors are known to contribute in the pathogenesis of melasma such as genetic predisposition, ultraviolet radiation, hormonal factors, oral contraceptives and drugs like phenytoin. Thyroid abnormalities were reported to occur with melasma. Skin pigmentation is a common manifestation in nutritional deficiencies and frequently associated with deficiency of vitamin B12 . Increased iron may affect the pattern and course of pigmentation, however it is unclear how they coexist. Vitamin D3 (cholecalciferol) is synthesized from 7-dehydrocholesterol by photochemical process in the skin and through successive hydroxylation to its active metabolite. 1, 25-dihydroxyvitamin D3 [1, 25(OH)2D3; calcitriol] is formed in liver and kidney. Intracellular receptor (VDR) helps in binding of vitamin D which helps the epithelial cells and melanocytes a target for vitamin D. Although vitamin D is used in the treatment of melanoma and psoriasis and active role of 1, 25(OH)2D3 in skin no reports of melasma associated with vitamin D reported. The dysfunction of 1,25(OH)2D3 - VDR system may lead to periodontal disease . Mineral bone density could be directly related to deficiency of vitamin D which also progress to osteoporosis. Studies have reported that anemia may predispose to periodontitis but the correlation was not determined. Until date, no studies reported any correlation or mere association between melasma, periodontitis and serum vitamin D abnormalities as well as decreased Hb levels. The present study was intended to assess the presence of periodontitis and vitamin D deficiency in melasma patients and evaluate clinical presence of periodontitis, which may occur in conjunction with melasma and vitamin D deficiency. The mere presence of melasma may help to investigate for further oral issues such as periodontitis and anemia which may or may not be associated with vitamin D abnormalities.

Patients visiting the Dept. of Oral medicine, with melasma on face within the age group of 30-70yrs in either gender were included in the study, matched with similar control group without melasma after obtaining informed consent.

The patients were divided into 2 groups. Group A, had Patients with melasma in whom 2 ml of blood was collected for estimation of serum-vitamin D levels, and complete blood picture was estimated for Haemoglobin percentage and clinical oral examination was evaluated for periodontitis. Group B served as control arm, where same procedure of blood parameter estimation and clinical examination protocol was followed as in group A.

Total number of 100 patients participated in the study, 50 in each group. The samples that resulted out of recruitment were tabulated and appropriate statistical analysis was done comparing the both groups with the presence or absence of periodontitis and serum vitamin D abnormalities and serum Hb% levels.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were patients with history of melasma and who were willing to be part of the study and patients who were not on any Systemic medication.

Exclusion Criteria:

* Exclusion criteria included patients who were not willing to be part of the study, patients who had endocrine disorders, patients with generalized pigmentation and as well as patients on steroid therapy.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total number of 100 patients participated in the study, 50 in each group. Patients visiting the Dept. of Oral medicine, with melasma on face within the age group of 30-70yrs in either gender were included in the study, matched with similar control group without melasma after obtaining informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Serum Vitamin D analysis | 3 -4 days
  I. The criteria for serum vitamin D analysis was followed which was laid by NATIONAL INSTITUTE OF HEALTH vitamin D fact sheet (2011) in both the groups using chemilumnescence method.
  <12 ng/ml -significant deficiency 12- 20 ng/ml - insufficiency >20 ng/ml - normal > 50 ng/ml - hypervitaminosis
Serum- hemoglobin levels | 1 day
  Evidence of pallor was checked clinically by examination of palpebral conjunctiva and correlated with serum haemoglobin percentage in both the groups using photometry method.
Clinical Periodontal index | 1 day
  The criteria to diagnose periodontitis clinically was followed by regulations laid down by Russell's periodontal index status , using mouth mirror and plain probe on all the gingival tissue circumscribing each tooth. It was assessed for gingival inflammation and periodontal involvement with loss of attachment. The evaluation was done by only one specialist.

CONTACTS AND LOCATIONS:
Overall Officials: NALLAN Ck CHAITANYA, mds, Principal Investigator — Panineeya Institute of dental sciences

IPD SHARING:
Plan to Share IPD: No